CLINICAL TRIAL: NCT04578340
Title: Long Term Outcomes Following Hernia Repair With Mesh
Status: Recruiting | Type: Observational
Sponsor: Endeavor Health (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Michael Ujiki MD, Director of Minimally Invasive Surgery; Chief, Division of Gastrointestinal and General Surgery, Endeavor Health
Other Study IDs: EH20-388
Record Dates: First submitted 2020-10-01; First posted 2020-10-08 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Abdominal Hernia
MeSH Terms: conditions — Hernia, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to establish the extent to which mesh improves quality of life and surgical outcomes following hernia repair.

DETAILED DESCRIPTION:
This is a large scale registry of prospectively collected medical record data and self-reported outcomes for those patients undergoing abdominal hernia repair with mesh.

ELIGIBILITY:
Inclusion Criteria:

* abdominal hernia repair using mesh

Exclusion Criteria:

* less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Multihospital system inclusive of all abdominal hernia repairs using mesh
Sampling Method: Non-Probability Sample
Enrollment: 4700 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Hernia recurrence rate | Within 5 years of initial hernia repair
  Should the hernia repair fail and the hernia reappears, this is counted as a recurrent hernia.
Patient quality of life | Up to 5 years postopertively
  Quality of life before and after surgery will be compared using various self-reported assessment tools/questionnaires.

SECONDARY OUTCOMES:
Postoperative infection rate | Up to 5 years postoperatively
  Infection related to hernia repair or mesh use will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- NorthShore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No